CLINICAL TRIAL: NCT03516799
Title: A Pilot Study of Acupuncture for Pain Management for AYA With Cancer
Brief Title: Acupuncture Intervention for AYA With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-014621
Record Dates: First submitted 2018-03-23; First posted 2018-05-04 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Palliative Care
Keywords: pain management of adolescent and young adults with cancer
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Non-randomized trial across four time points at one study site
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (ACU) Group (Experimental): The group of participants who opt in to acupuncture
  Interventions: Other: Acupuncture
- Treatment-as-Usual (TAU) Group (No Intervention): The group of participants who enroll in the study but opt out of acupuncture (treatment-as-usual)

INTERVENTIONS:
Other: Acupuncture — Acupuncture is a method of Traditional Chinese Medicine that consists of the insertion of thin, sterile, FDA-approved disposable needles on specific acupuncture points (acupoints).
  Arms: Acupuncture (ACU) Group

SUMMARY:
The aim of the study is to innovatively extend acupuncture research in adult oncology to adolescents and young adults (AYA) by piloting a tailored acupuncture protocol for pain management in AYA in the Children's Hospital of Philadelphia (CHOP's) Center for Integrative Health.

DETAILED DESCRIPTION:
Acupuncture is an integrative medicine (IM) with a growing evidence base that is often incorporated into comprehensive pain management in adult oncology. However, it is under-utilized and under-researched in pediatric oncology, especially with adolescents and young adults (AYA). Acupuncture is a promising palliative therapy to manage pain and improve quality of life (QOL) of AYA. AYA are underserved and typically endure more morbidity and longer treatments than younger patients. More than half report at least three debilitating cancer-related symptoms and their QOL is significantly lower compared to norms, with symptoms being the greatest contributor to poor QOL. Not surprisingly, AYA identify pain management as an unmet need, leading a majority of AYA to want information on IM or seek it for treatment. Given the potential benefit of acupuncture for addressing unmet needs of AYA by reducing physical suffering, and the established difficulty with pain management using conventional methods, there is a critical need to establish the efficacy of acupuncture for pain management in AYA. The few studies that have evaluated acupuncture in pediatric oncology, demonstrating it to be safe, accepted, and associated with symptom relief are uncontrolled, retrospective, and/or unprotocolized, and none focus on AYA. To establish the evidence base for acupuncture in AYA oncology, research is needed to determine and test optimal acupuncture protocols.

ELIGIBILITY:
AYA Inclusion Criteria:

* Report a pain severity score of ≥ 4 in last 7 days on an 11-point (0-10) numerical rating scale and reports a pain distress score of ≥ 2 on a 5-point numerical rating scale
* Males or females age 13 to 24 years
* On treatment for cancer for at least one month or within two years of completing treatment
* Not expected to be terminal within the next 6 months
* Absence of infection or bleeding disorder
* Physically and medically able to get to the acupuncture clinic
* Able to read and write English

AYA Exclusion Criteria:

* Absence of inclusion criteria above
* Parents'guardians or subjects who, in the opinion of the investigator, may be non-compliant with the study schedules or procedures
* Cognitive impairments that would limit AYA's ability to complete measures or to independently care for health as determined by medical team

Parent/Guardian Inclusion Criteria:

* Be primary parent/guardian of the AYA participant
* Be able to read and write English

Parent/Guardian Exclusion Criteria:

* Cognitive impairments that would limit the parent/guardian's ability to complete measures
* Absence of inclusion criteria above

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Acceptability of use of Acupuncture for pain management of AYA and associates | 15 weeks
  Number of participants who report satisfaction and intention for future use through a qualitative semi-structured interview. ("How satisfied were you with the number of acupuncture sessions you received over the course of the study?"...."how likely would you be to continue to receive acupuncture in the future?")
Number of acupuncture sessions completed | 15 weeks
  Number of sessions participants complete and time between sessions, which will be logged by research team for feasibility.
Number of participant-reported barriers to participating in acupuncture sessions for AYA who opt in | 15 weeks
  Number of participants who report barriers to participation during qualitative semi-structured interview for feasibility. ("How difficult or inconvenient did you find going to your acupuncture appointment over the course of these past 10 weeks to be?")
Incidence of patient-reported adverse events of AYA who opt in to acupuncture relative to those who opt out | 15 weeks
  Limited report of acupuncture-related side effects which will be logged as patient reported outcomes ("did you experience any adverse events?") post-acupuncture sessions. Treatment-Related Adverse Events as Assessed by CTCAE v4.0, change from baseline in pain scores.

SECONDARY OUTCOMES:
Acupuncture as a pain management tool | 15 weeks
  To determine the preliminary efficacy of acupuncture for pain management of AYA. Compared to AYA who opt out, AYA who receive acupuncture will report, from baseline to post-treatment: reduced severity of pain, improvement in QOL, reduced pain interference, and symptom-related distress through a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Schwartz, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No